CLINICAL TRIAL: NCT00453947
Title: Non Invasive Positive Airway Pressure And Risk Of Myocardial Infarction In Acute Cardiogenic Pulmonary Edema: Continuous Positive Airway Pressure Vs Non Invasive Positive Pressure Ventilation
Brief Title: Non-Invasive Ventilation in Pulmonary Edema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ospedale S. Giovanni Bosco (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: gbosco2
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Last update posted 2007-03-29 (Estimated); Status verified 2007-03

CONDITIONS: Pulmonary Edema; Myocardial Infarction
MeSH Terms: conditions — Pulmonary Edema; Myocardial Infarction | interventions — Continuous Positive Airway Pressure; Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: CPAP and Non Invasive Ventilation

SUMMARY:
This randomized controlled trial is primarily aimed at assessing the rate of acute myocardial infarction with the two noninvasive ventilatory techniques, non-invasive intermittent positive pressure ventilation and non-invasive continuous positive airway pressure.

DETAILED DESCRIPTION:
Objective: To determine whether the application of non-invasive intermittent positive pressure ventilation (n-IPPV) increases the incidence of acute myocardial infarction (AMI) in patients with acute respiratory failure (ARF) secondary to acute cardiogenic pulmonary edema (ACPE), as opposed to non-invasive continuous positive airway pressure (n-CPAP).

Background Both n-CPAP or n-IPPV are used to treat ACPE complicated by ARF. Two previous studies, however, report an increased rate of AMI associated with the use of n-IPPV.

Methods: Fifty-two patients with severe ARF consequent to ACPE were randomized to receive n-CPAP (n=27) or n-IPPV (n=25), both associated with standard medical therapy. Cardiac markers, electrocardiogram and clinical-physiological parameters were monitored at study entry, after 30 and 60 minutes, and every 6 hours for the first two days.

ELIGIBILITY:
Inclusion Criteria:

* rapid onset of the symptoms
* severe dyspnoea at rest
* respiratory rate > 30 breaths per minute
* use of accessory respiratory muscles
* oxygen saturation (SpO2) inferior to 90% with an inspiratory oxygen fraction of 60% via a Venturi mask
* radiological findings of ACPE

Exclusion Criteria:

* acute ischemic heart disease (myocardial infarction, chest pain, ST elevation)
* hemodynamic instability (i.e. systolic blood pressure < 90 with dopamine or dobutamine infusion ≥ 5 mcgr/Kg/min) or life-threatening arrhythmias
* need for immediate endotracheal intubation (respiratory arrest, bradypnea or gasping)
* inability to protect the airways
* impaired sensorium (i.e. unconsciousness or agitation)
* inability to clear secretions
* respiratory tract infection
* recent oesophageal/gastric surgery
* gastrointestinal bleeding
* facial deformities
* hematological malignancy or cancer with an Eastern Cooperative Oncology Group performance status ≥ 2
* chronic respiratory failure necessitating long-term oxygen therapy
* diagnosis of myocardial infarction, pulmonary embolism, pneumonia, exacerbation of chronic obstructive pulmonary disease, pneumothorax in the previous 3 months
* denial or refusal of intubation
* claustrophobia
* inclusion in other research protocols

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-07; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
The rate of Acute Myocardial Infarction

SECONDARY OUTCOMES:
Rate of endotracheal intubation
Mortality
Time of recovery (i.e. duration of ventilatory assistance)
High Dependency Unit and hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Ferrari, MD, Principal Investigator — Ospedale San Giovanni Bosco ASL4 Torino Italy
Locations (1):
- Ospedale San Giovanni Bosco Medicina d'Urgenza, Torino, Torino, Italy

REFERENCES:
- [Derived] Ferrari G, Olliveri F, De Filippi G, Milan A, Apra F, Boccuzzi A, Converso M, Navalesi P. Noninvasive positive airway pressure and risk of myocardial infarction in acute cardiogenic pulmonary edema: continuous positive airway pressure vs noninvasive positive pressure ventilation. Chest. 2007 Dec;132(6):1804-9. doi: 10.1378/chest.07-1058. Epub 2007 Oct 1. PMID 17908705